CLINICAL TRIAL: NCT07115589
Title: Impacts of Home-based Cardiovascular Rehabilitation on the Physical Fitness of Children, Adolescents and Young Adults With Congenital Heart Disease: the "Muscle Your Heart" Program
Brief Title: Home-based Cardiovascular Rehabilitation in Young Patients With Congenital Heart Disease: the "Muscle Your Heart" Program
Acronym: Muscletoncoeur
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2024/23; 2024-A01806-41 (Other: ID-RCB number)
Record Dates: First submitted 2025-06-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: CHD - Congenital Heart Disease
Keywords: Congenital heart disease; Paediatric; Cardiovascular rehabilitation; Adapted physical activity; Therapeutic patient education
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fully home-based cardiovascular rehabilitation program (Experimental): 3-month cardiovascular rehabilitation program entirely at home, combining adapted physical activity, therapeutic education and psychosocial support
  Interventions: Other: Muscle Your Heart home-based program

INTERVENTIONS:
Other: Muscle Your Heart home-based program — 2 one-hour sessions of adapted physical activity per week - HIIT and free adapted physical activity - 1 one-hour monthly therapeutic patient education session - A dedicated platform - Adapted physical activity educators - Dedicated education therapeutic nurses

SUMMARY:
Standard cardiovascular rehabilitation is performed in a medical care and rehabilitation centre. However, it may not be adapted to the patient's profile and there are few medical care and rehabilitation centres specialized in pediatric cardiology. The objective of this study is to evaluate the impact of cardiovascular rehabilitation entirely at home on the physical fitness of young patients with congenital heart disease.

DETAILED DESCRIPTION:
Young patients with congenital heart disease suffer from physical deconditioning [1], negatively impacting the quality of life [2, 3], due in particular to obstacles stated by the patient's social environment [4, 5]. For this, there is cardiovascular rehabilitation, however, it may not be adapted to the patient's profile and there are few specialized centres in France. In the sense, the QUALIREHAB program, tested in a randomized controlled trial, was created. This 3-month hybrid program (at the patient's home and in a medical care and rehabilitation centre), combining adapted physical activity, patient therapeutic education and psychosocial support, has demonstrated positive effects on quality of life, level of physical activity, knowledge of the disease, body mass index and mental health [6].

However, this program has limitations, including the need for a medical care and rehabilitation centre near the patient's home.

This study, evaluating the impact of a 3-month cardiovascular rehabilitation program entirely at home, will improve this program by taking into account its limitations and will apply it to real life, without all the human, financial and material resources of a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Indication for home cardiovascular rehabilitation given by the referring cardiologist as part of routine care.
* Follow-up for congenital heart disease in the ACC-CHD classification.
* Patient aged 8 to 25 years at the time of inclusion.
* Consent of the adult patient or the parents or legal guardians of the minor patient.
* Social security affiliation (excluding AME).
* VO2max and/or SV1 < -1.64 z-score for patients aged 8 to 17 years or VO2max < 80% and/or SV1 < 55% of theoretical VO2max for patients aged 18 to 25 years

Exclusion Criteria:

* Unstable and/or severe heart failure: severe heart failure (NYHA functional class IV), recent decompensated heart failure requiring hospitalisation and/or any significant change in medication (< 3 months before inclusion), systolic ventricle dysfunction (left ventricular or systemic ventricular ejection fraction < 50%).
* Severe hypoxemia: pulse oxygen saturation (SpO2) at rest < 85%, and/or SpO2 at exercise < 80%, and/or patient requiring oxygen therapy.
* Pulmonary hypertension as defined by the 2020 ESC guidelines, whatever the aetiology.
* Significant systolic right ventricle (sRV) hypertension (Srv pressure > 50% of systemic systolic pressure).
* Uncontrolled arrhythmia: symptomatic arrhythmia treated or untreated at rest and/or during exercise, treated arrhythmia with sustained supraventricular or ventricular tachycardia on ECG monitoring or during exercise and/or CPET, occurrence or aggravation of any supraventricular or ventricular arrhythmia during exercise and/or CPET.
* Advanced atrioventricular block (degree 2 or 3), occurrence or aggravation of any conduction disorder during exercise and/or CPET.
* Uncontrolled arterial hypertension at rest (blood pressure at rest during the consultation > 140/90 mmHg in adults, > 95th percentile in children).
* Acute or recent myocarditis and pericarditis (< 3 months).
* Symptomatic aortic or subaortic stenosis (mean gradient > 50 mmHg).
* Non-corrected coarctation of the aorta (surgical or catheter-based repair) with a clinical systolic gradient > 20 mmHg.
* Dilatation of the aorta (aortic root > 40 mm in adults, > 2 z-score in children) (http://www.parameterz.com/sites/aortic-root) except in the case of repaired CHD with dilatation of the aorta inherent in the malformation and without risk of aortic dissection (tetralogy of Fallot, transposition of the great vessels, pulmonary atresia IVC, common trunk artery).
* Severe obstructive hypertrophic cardiomyopathy.
* Acute systemic disease.
* Recent intracardiac thrombus (< 3 months), embolism or thrombophlebitis.
* Inability to follow instructions and/or home rehabilitation and/or answer questionnaires, as determined by the investigator.
* Absolute contraindications for CPET: fever, uncontrolled asthma, respiratory failure, acute myocarditis or pericarditis, uncontrolled arrhythmias causing symptoms or hemodynamic compromise, uncontrolled heart failure, acute pulmonary embolus or pulmonary infarction, and patients with mental impairment leading to inability to cooperate.
* Inability to undergo the physical intervention: inability to physically exercise, any invasive medical intervention occurring within 6 months preceding the inclusion or scheduled during the 3-month study period (such as cardiac surgery, catheter-based intervention, orthopedic surgery, chemotherapy for cancer, or any other significant medical treatment or intervention, as determined by the investigator).
* For female patients: pregnancy, planning to become pregnant, or breastfeeding woman following questioning of the patient.
* Any other clinical and/or pharmacological treatment that is believed to interfere with the study or the optimal clinical care.
* Patients deprived of their liberty due to ongoing legal procedure, adult patients under guardianship or curatorship, or unable to personally express their consent.
* Patients who have benefited from cardiovascular rehabilitation in the 12 months preceding inclusion.
* Patient participating or wishing to participate in any interventional clinical research (drug trial, medical device, non-drug trial).

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of the maximal oxygen consumption (VO2max) obtained in the cardiopulmonary exercise test (CPET) | baseline and at the end of the 3-month program (week 12)

SECONDARY OUTCOMES:
First ventilatory anaerobic threshold obtained at the CPET | at week 0 and at week 14 (last visit after the end of the rehabilitation program)
Ventilatory efficiency (VE/VCO2 slope) obtained at the CPET | at week 0 and at week 14 (last visit after the end of the rehabilitation program)
Maximum oxygen pulse obtained at the CPET | at week 0 and at week 14 (last visit after the end of the rehabilitation program)
Maximum workload in watt obtained at the CPET | at week 0 and at week 14 (last visit after the end of the rehabilitation program)
Quality of life assessed with Pediatric Quality of Life questionnaire (PedsQL) questionnaire (self and proxy) | at week 0 and at week 14
  This is a validated questionnaire for patients aged between 2 and 25, comprising 23 items covering 4 different areas: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and academic functioning (5 items). The proxy questionnaire, designed for parents and those close to the child, assesses parents' perceptions of the quality of life associated with their child's state of health. Each item is scored from 0, when there is no problem, to 4, when there is always a problem.
Level of physical activity assessed with questionnaires for 8 to 17-year-old | at week 0 and at week 13
  The questionnaire for children aged 8 to 17 years included is the CAPAS-Q (Children and adolescents physical activity and sedentary questionnaire). The CAPAS-Q was developed as a clinical and field tool to provide indicators of physical activity and sedentary behaviour. The CAPAS-Q allows indicators such as the duration and intensity of physical activity to be addressed in different contexts (school, outside school, sports and leisure activities, transport). Physical activity is scored from 1 (inactive) to 4 (very active) and sedentary lifestyle is scored from 1 (not sedentary, active enough) from 6 (sedentary).
Level of physical activity assessed with questionnaires for over 18-year-old | at week 0 and at week 13
  For patients over 18 years of age, the short version of the IPAQ (International physical activity questionnaire) was chosen. This questionnaire assesses overall physical activity and sedentary behaviour over the last 7 days. The questionnaire looks at vigorous and moderate activity, walking, and time spent sitting (sedentary lifestyle), whether during leisure activities, at work, in daily life or on public transport. The questionnaire classifies the subject according to 3 levels of activity: inactive, moderate, high.
Level of physical activity assessed with accelerometers and questionnaires | at week 0 and at week 13
  Patients will wear an accelerometer for 7 days, to objectively measure their level of physical activity. This tool must be removed during aquatic activities or during activities involving physical contact.
Muscle strength of the upper limbs assessed by handgrip test | at week 0 and at week 14
  The Handgrip test consists of squeezing the handle of a hand dynamometer. The patient chooses their preferred hand and squeezes the handle as hard as they can for 3 seconds. The task was repeated 3 times, with 30 seconds rest between trials. The best trial is used as an indicator of maximum upper limb strength.
Muscle strength of lower limbs assessed Standing long jump test | at week 0 and at week 14
  For the lower limbs, the Standing long jump test is used. The patient stands with feet together and jumps forward as far as possible. After the jump, the patient must remain motionless with both feet on the ground. If he loses his balance or touches an object, he must repeat the jump. The distance between the jump line and the heels is measured. The patient performs 2 trials, the longest distance being used as an indicator of maximum lower limb strength.

CONTACTS AND LOCATIONS:
Overall Officials: Pr Pascal AMEDRO, MD,PhD, Study Director — CHU de Bordeaux - Hôpital Cardiologique Haut Lévêque
Locations (1):
- CHU de Bordeaux - Hôpital Cardiologique Haut Lévêque, Pessac, France, France

REFERENCES:
- See also: Amedro, P., Gavotto, A., Guillaumont, S., Bertet, H., Vincenti, M., De La Villeon, G., et al. (2018). Cardiopulmonary fitness in children with congenital heart diseases versus healthy children. Heart (British Cardiac Society), 104(12), 1026-1036. — https://doi.org/10.1136/heartjnl-2017-312339
- See also: Amedro, P., Dorka, R., Moniotte, S., Guillaumont, S., Fraisse, A., Kreitmann, B., et al. (2015). Quality of Life of Children with Congenital Heart Diseases: A Multicenter Controlled Cross-Sectional Study. Pediatric cardiology, 36(8), 1588-1601. — https://doi.org/10.1007/s00246-015-1201-x
- See also: Amedro, P., Picot, M. C., Moniotte, S., Dorka, R., Bertet, H., Guillaumont, S., et al. (2016). Correlation between cardio-pulmonary exercise test variables and health-related quality of life among children with congenital heart diseases. International — https://doi.org/10.1016/j.ijcard.2015.11.028
- See also: Longmuir, P. E., & McCrindle, B. W. (2009). Physical activity restrictions for children after the Fontan operation: disagreement between parent, cardiologist, and medical record reports. American heart journal, 157(5), 853-859 — https://doi.org/10.1016/j.ahj.2009.02.014
- See also: Swan, L., & Hillis, W. S. (2000). Exercise prescription in adults with congenital heart disease: a long way to go. Heart (British Cardiac Society), 83(6), 685-687 — https://doi.org/10.1136/heart.83.6.685
- See also: Craig, C. L., Marshall, A. L., Sjöström, M., Bauman, A. E., Booth, M. L., Ainsworth, B. E., Pratt, M., et al. (2003). International physical activity questionnaire: 12-country reliability and validity. Medicine and science in sports and exercise, 35(8 — https://doi.org/10.1249/01.MSS.0000078924.61453.FB
- See also: Hagströmer, M., Oja, P., & Sjöström, M. (2006). The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public health nutrition, 9(6), 755-762 — https://doi.org/10.1079/phn2005898
- See also: Wind, A. E., Takken, T., Helders, P. J., & Engelbert, R. H. (2010). Is grip strength a predictor for total muscle strength in healthy children, adolescents, and young adults?. European journal of pediatrics, 169(3), 281-287 — https://doi.org/10.1007/s00431-009-1010-4
- See also: Castro-Piñero, J., Ortega, F. B., Artero, E. G., Girela-Rejón, M. J., Mora, J., Sjöström, M., & Ruiz, J. R. (2010). Assessing muscular strength in youth: usefulness of standing long jump as a general index of muscular fitness. Journal of strength and — https://doi.org/10.1519/JSC.0b013e3181ddb03d